CLINICAL TRIAL: NCT00894101
Title: A Phase II/III, Open Label, Non-Randomized, Multi-Center Study of Positron Emission Tomography Imaging With [F-18] FLT Compared to [F-18] FDG in Cancer Patients for Treatment Evaluation
Brief Title: Positron Emission Tomography Imaging With [F-18] FLT Compared to [F-18] FDG in Cancer Patients for Treatment Evaluation
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The main sponsor of this multi-center trial has submitted this protocol. A single participating site should not register this study.
Sponsor: University of California, Irvine (Other)
Responsible Party: Dr. Orhan Nalcioglu, Professor & Director, University of California, Irvine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS# 2009-6857
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — alovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [F-18] FLT and FDG (Experimental)
  Interventions: Drug: [F-18] FLT

INTERVENTIONS:
Drug: [F-18] FLT — 10 mCi [F-18] FLT and 10 mCi [F-18] FDG will be used for PET imaging.

SUMMARY:
The purpose of this study is to investigate the clinical value of serial quantitative [F-18] FLT as a PET imaging tool in head and neck cancer patients clinically scheduled with radiation or radiation-chemotherapy combination in terms of safety and efficacy. Standard [F-18] FDG PET will be the active comparator.

ELIGIBILITY:
Inclusion Criteria:

1. Patient provides written Informed Consent and is willing to comply with protocol requirements
2. Patient is at least 18 years of age on the day of dosing (male or female of any race or ethnicity)
3. Patient is capable of lying still in the PET scanner for the protocol required time frame(s)
4. Patient has a diagnosis of one of the following malignancies (TNM Staging System):

   * Lung cancer (T3 grade up, node positive, but no metastatic disease)
   * Head and neck cancer (T3 grade up, node positive, but no metastatic disease)
5. Patient has undergone a comparative, diagnostic procedure with lesion(s) visible, other than ultrasound, that includes, but is not limited to computed tomography (CT), magnetic resonance imaging (MRI), nuclear medicine imaging, endoscopy, laparoscopy, standard abdominal x-ray, biopsy and/or surgery for one of the above mentioned areas
6. Patient is scheduled to start radiotherapy or a chemoradiotherapy regimen for curative intent
7. As a part of his/her standard radiotherapy or chemoradiotherapy regimen, patient is scheduled to have clinical [F-18] FDG PET scans pre treatment and post treatment (at about 4 weeks (±1 week) after the start of therapy)
8. Patient is scheduled to have the investigational, pre treatment [F-18] FLT PET scan recommended to be within ± 2 days of the clinical, pre treatment [F-18] FDG PET scan
9. Patient has not received or intends to receive 5-fluorouracil (5-FU-chemotherapeutic agent)
10. Patient has a score of greater than or equal to (≥) 60% on the Karnofsky Performance Status Scale

Exclusion Criteria:

Exclude a patient from this study if the patient does not fulfill the inclusion criteria, or if any of the following conditions are observed:

1. Patient is a pregnant or lactating female. These methods will be used to exclude the possibility of pregnancy:

   * by testing on site at the institution (serum or urine βHCG) within 48 hours prior to the start of each investigational product administration,
   * by surgical history (eg, tubal ligation or hysterectomy),
   * by patient's history of being post menopausal with a minimum 1 year without menses.
2. Patient is undergoing treatment with palliative intent
3. Patient has received an investigational compound and/or medical device within 14 days before admission into this study
4. Patient has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post-dose follow-up examinations
5. Patient is determined by the Investigator that he/she is clinically unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
The basic safety data of [F-18] FLT tracer will be collected. The treatment response evaluated based on the [F-18] FLT results will be compared to the response evaluated based on the standard PET trace [F-18] FDG. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, UCI Medical Center, Orange, California, United States